CLINICAL TRIAL: NCT02707757
Title: Predictors of Response to Treatment With Iron and Erythropoietin in Dialysis Anaemia
Brief Title: Treatment Response in Dialysis Anaemia
Acronym: PRIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14HH1987
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Anaemia; Haemodialysis
Keywords: Haemodialysis; Anaemia; Iron; Erythropoeitin stimulating agents
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron sucrose (Active Comparator): Iron sucrose 200mg for 5 doses
  Interventions: Drug: Iron sucrose
- Neorecormon (Active Comparator): Incremental increase in dose along following parameters: 1000-2000-3000-4000-6000-8000-12000
  Interventions: Drug: Erythopoietin stimulating agent

INTERVENTIONS:
Drug: Iron sucrose — 1gram of iron sucrose (5 200mg aliquots) administered if participant's haemoglobin is less than 9.5g/dl
  Other Names: Venofer
  Arms: Iron sucrose
Drug: Erythopoietin stimulating agent — Incremental increase in dose of erythropoeitin stimulating agent being administered as per a pre-defined criteria
  Other Names: Neorecormon
  Arms: Neorecormon

SUMMARY:
Anaemia in dialysis patients requires treatment with frequent dose adjustments. There are two current possible treatments for anaemia which are iron and erythropoietin stimulating agents (ESA). Dosages of these medications are currently guided by a patient's ferritin levels and haemoglobin, but these markers are known to be inaccurate. The current clinical protocol therefore tends towards overuse of both agents which can be associated with toxicity, and the reliance on these markers prevents retrospective assessment of treatment responsiveness. This study is designed to investigate the factors which predict which agent would produce a better response. Patients with a fall in haemoglobin will be given treatment with either iron or an increased dose of ESA as they are currently, but allocated at random rather than by poorly performing biochemical markers. The iron treated and ESA treated groups can then be analysed for factors which predict response in o

ELIGIBILITY:
Inclusion Criteria:

* All prevalent haemodialysis patients of the Imperial Renal and Transplant Centre will be eligible for inclusion if they have been on dialysis for more than 3 months

Exclusion Criteria:

* Patients with a bone marrow disorder, active infection or active malignancy will be excluded as these are non-renal causes of anaemia. Patients unable to give informed consent will also not be included within the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Dr Ashby, MBBS, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (2):
- United Kingdom (2):
  - Imperial Renal and Transplant Centre, London
  - Imperial NHS Healthcare Trust, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 197 prevalent haemodialysis patients
Pre-assignment Details: Recruitment from the study was the prevalent haemodialysis population. Those whom were recruited (197) were then followed until the monthly Hb, taken within routine haemodialysis care, triggered a randomisation event.
  Exclusion criteria for either recruitment or a randomisation event:
  Overt blood loss Haematological or other malignancy
Period: Overall Study
Arm/Group | Iron Sucrose | Neorecormon
Started (This refers to the number of times to which a participant was allocated to each respective treatment. A participant could be re-randomised 6 months following initial randomisation. Not all participants were randomised due to not meeting randomisation criteria.) | 88 | 96
Completed | 76 | 84
Not Completed | 12 | 12
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 1
Not completed — Adverse Event | 6 | 4
Not completed — Renal transplant/elective operation | 1 | 5

BASELINE CHARACTERISTICS:
Population: Analysed on a per protocol rather than intention to treat basis
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Sucrose | Neorecormon | Total
Number analyzed (Participants) | 76 | 84 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 78
  >=65 years | 39 | 43 | 82
Age, Continuous [Mean (Full Range); unit: years] | 63.22 [31 to 86] | 63.10 [25 to 91] | 63.16 [25 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 54 | 60 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 34 | 41 | 75
  Ethnicity: Asian | 31 | 28 | 59
  Ethnicity: Black | 9 | 12 | 21
  Ethnicity: Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 76 | 84 | 160

OUTCOME MEASURES:

1. Primary Outcome: Haemoglobin Increase of Greater or Equal to 5g/l Following Receipt of Treatment
Time Frame: 2 months
Population: Per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Sucrose | Neorecormon
Number analyzed (Participants) | 76 | 84
Participants | 53 | 61

ADVERSE EVENTS:
Arm/Group | Iron Sucrose | Neorecormon
All-Cause Mortality (participants affected / at risk) | 3/88 | 2/96
Serious Adverse Events (participants affected / at risk) | 17/88 | 21/96
Other Adverse Events (participants affected / at risk) | 2/88 | 1/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iron Sucrose (N=88) | Neorecormon (N=96)
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Cardiac arrhythmia (Cardiac disorders) | 1 | 2
Bacteraemia (Infections and infestations) | 1 | 2
Soft tissue infection (Skin and subcutaneous tissue disorders) | 3 | 0
Cervical discitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Vasculitis (Immune system disorders) | 0 | 1
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Psoas abscess (Infections and infestations) | 1 | 1
Stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iron Sucrose (N=88) | Neorecormon (N=96)
Transfusion (Blood and lymphatic system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes